CLINICAL TRIAL: NCT01545271
Title: Xenon and Cooling Therapy in Babies at High Risk of Brain Injury Following Poor Condition at Birth: A Randomised Pilot Study
Brief Title: Xenon and Cooling Therapy in Babies at High Risk of Brain Injury Following Poor Condition at Birth
Acronym: CoolXenon2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH/2011/3799; 2011-005397-34 (EudraCT Number); 12/SW/0010 (Other: NRES Committee South West)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Hypoxic Ischaemic Encephalopathy
Keywords: Xenon; Hypothermia; Hypoxic Ischemic Encephalopathy; Newborn; Term; Neuroprotection; Cooling; HIE
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 72h cooling + 18h xenon inhalation (Experimental): Babies in poor condition at birth and referred to our neonatal unit for standard therapy of cooling to 33.5 degree C body temperature will be randomised to receive xenon gas at 50% concentration for 18 hours
  Interventions: Drug: xenon gas; Device: Whole body cooling
- Standard 72 h whole body cooling therapy (Active Comparator): Whole body cooling therapy to rectal temperature of 33.5 degree Centigrade (standard therapy)
  Interventions: Device: Whole body cooling

INTERVENTIONS:
Drug: xenon gas — Inhalation via endotracheal tube of 50% xenon for 18 hours, including during transport for outborn babies, starting within 5 hours after birth.
  Other Names: LENOXe
  Arms: 72h cooling + 18h xenon inhalation
Device: Whole body cooling — Cooling of baby to reduce rectal temperature to 33.5 degree Centigrade(standard treatment), including during transport for outborn babies, starting within 3 hours after birth.

SUMMARY:
This study examines the effect of inhaled xenon gas in the treatment of newborn infants with hypoxic-ischemic encephalopathy (HIE) in combination with cooling, which is the standard treatment for this condition. The hypothesis is that the xenon + cooling combination will produce better neuroprotection than the standard treatment of cooling alone.

ELIGIBILITY:
Infants will be eligible for for the trial if the St Michael's hospital standard inclusion criteria for cooling and additional inclusion criteria for xenon administration are met.

St Michael's hospital standard inclusion criteria for standard hypothermia treatment of 72 hrs:

A: Neonates born at greater than 36 weeks gestation (estimated or clinical assessment) with at least ONE of the following:

1. Apgar score of ≤5 at ten minutes after birth
2. Continued need for resuscitation, including tracheal or mask ventilation, at ten minutes after birth
3. Acidosis, defined as either umbilical cord pH or any arterial, venous or capillary pH within 60 minutes of birth less < 7.00
4. Base deficit ≥16 mmol/L in umbilical cord blood sample or any blood sample within 60 minutes of birth (arterial or venous blood).

If the infant meets criterion A then assess for neurological abnormality using criterion B and C (by trained personnel):

B: Moderate or Severe encephalopathy as evidenced by any of the following:

1. Altered state of consciousness (reduced or absent responses or pathological irritability and hyper responsive and at least ONE or more of the following:
2. Hypotonia
3. Abnormal reflexes including oculomotor or pupillary abnormalities
4. Absent or weak suck
5. Clinical seizures, as recorded by trained personnel

And

C: At least 30 minutes duration of amplitude-integrated electroencephalography (aEEG) recording that shows abnormal background aEEG activity. The decision to cool is based on the worst 30 min section of the aEEG, not the best [35] or seizures (clinical or electrical) thus meeting ONE of the following:

1. Normal background with some (> 5 min) electrical seizure activity
2. Moderately abnormal activity (upper margin of trace >10μV and lower margin <5μV)
3. Suppressed activity (upper margin of trace <10μV and lower margin of trace <5μV)
4. Definite seizure activity

Additional inclusion criteria for xenon:

Before being considered for additional inhaled xenon therapy via the breathing gas mixture, the infant would need to meet further additional entry criteria (all must be met):

1. Intubated, ventilated, sedated, being cooled
2. ≤ 5 hours old
3. Any seizures under control
4. Weight > 2nd centile for gestational age
5. Stable cardiovascular parameters; Mean arterial pressure >40mmHg.
6. Oxygen requirement via mechanical ventilator ≤ 40%.
7. Positive End Expiratory Pressure (PEEP) requirement ≤ 6cm H2O
8. Arterial pCO2 within acceptable range (<7kPa)
9. Absence of major congenital abnormalities, imperforate anus and in particular any bowel obstruction, congenital abnormalities suggestive of chromosomal anomaly or other syndromes that include brain dysgenesis. Congenital syndromes affecting the brain should be excluded when diagnosed.

Exclusion criteria for cooling in the CoolXenon2 study

1. Infants expected to be greater than 3 hours of age at the time of starting cooling treatment.
2. Futility. Where prognosis is considered to be hopeless e.g. no cardiac output for 20 minutes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Death and moderate or severe disability - Bayley III | at 18 months of age
  Bayley Scales of Infant and Toddler Development III (Bayley III) has three domains: cognition, language and motor skills. Each domain is based on a series of examinations of different severity. The lower cut off level is 55 for cognition, 47 for language and 46 for motor. The upper value can be 145. Assessment of hearing and vision: severe hearing loss defined as inability to hear without amplification; severe visual loss defined as being unable to move independently.

SECONDARY OUTCOMES:
Brain MRI | less than 2 weeks of age
  Magnetic Resonance Imaging findings at less than 2 weeks of age
Amplitude Integrated Electroencephalogram (aEEG) grading | Before hospital discharge; usually within one week of birth
  Number of hours after birth when aEEG voltage has reached a normal or discontinuous normal pattern

OTHER OUTCOMES:
Number of normal infants | 18-24 months
  Bayley III composite score ≥ 85 and no neurosensory disability as described above

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Thoresen, Professor, Principal Investigator — University of Bristol
Locations (1):
- St Michael's Hospital, Bristol, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chakkarapani E, Thoresen M, Hobbs CE, Aquilina K, Liu X, Dingley J. A closed-circuit neonatal xenon delivery system: a technical and practical neuroprotection feasibility study in newborn pigs. Anesth Analg. 2009 Aug;109(2):451-60. doi: 10.1213/ane.0b013e3181aa9550. PMID 19608817
- [Background] Hobbs C, Thoresen M, Tucker A, Aquilina K, Chakkarapani E, Dingley J. Xenon and hypothermia combine additively, offering long-term functional and histopathologic neuroprotection after neonatal hypoxia/ischemia. Stroke. 2008 Apr;39(4):1307-13. doi: 10.1161/STROKEAHA.107.499822. Epub 2008 Feb 28. PMID 18309163
- [Background] Thoresen M, Hobbs CE, Wood T, Chakkarapani E, Dingley J. Cooling combined with immediate or delayed xenon inhalation provides equivalent long-term neuroprotection after neonatal hypoxia-ischemia. J Cereb Blood Flow Metab. 2009 Apr;29(4):707-14. doi: 10.1038/jcbfm.2008.163. Epub 2009 Jan 14. PMID 19142190
- [Background] Chakkarapani E, Dingley J, Liu X, Hoque N, Aquilina K, Porter H, Thoresen M. Xenon enhances hypothermic neuroprotection in asphyxiated newborn pigs. Ann Neurol. 2010 Sep;68(3):330-41. doi: 10.1002/ana.22016. PMID 20658563
- [Background] Chakkarapani E, Thoresen M, Liu X, Walloe L, Dingley J. Xenon offers stable haemodynamics independent of induced hypothermia after hypoxia-ischaemia in newborn pigs. Intensive Care Med. 2012 Feb;38(2):316-23. doi: 10.1007/s00134-011-2442-7. Epub 2011 Dec 13. PMID 22160201
- [Derived] Dingley J, Liu X, Gill H, Smit E, Sabir H, Tooley J, Chakkarapani E, Windsor D, Thoresen M. The feasibility of using a portable xenon delivery device to permit earlier xenon ventilation with therapeutic cooling of neonates during ambulance retrieval. Anesth Analg. 2015 Jun;120(6):1331-6. doi: 10.1213/ANE.0000000000000693. PMID 25794112
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452

DOCUMENTS (1):
  • Study Protocol (2013-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT01545271/Prot_000.pdf